CLINICAL TRIAL: NCT01160055
Title: Identification and Characterisation of the Bacteria Causing Acute Otitis Media (AOM) Episodes in Young Children in Egypt
Brief Title: Study to Characterize and Identify Bacteria Causing Acute Otitis Media in Young Egyptian Children
Status: Withdrawn | Type: Observational
Why Stopped: Key aspects linked to sample management and analysis were not met during feasibility assessment limiting the ability of the study to reach its objectives.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113368
Record Dates: First submitted 2010-07-01; First posted 2010-07-12 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Infections, Streptococcal
MeSH Terms: conditions — Streptococcal Infections | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Middle ear fluid, Urine.

GROUPS / COHORTS (2):
- Cohort A: Subjects with a new episode of Acute Otitis Media (<3 days of onset) who have not yet received antibiotic therapy for the episode.
  Interventions: Procedure: Middle ear fluid and urine.
- Cohort B: Subjects who have had a diagnosis of Acute Otitis Media within 2-3 days prior to study enrolment and received antibiotic therapy, but remain symptomatic.
  Interventions: Procedure: Middle ear fluid and urine.

INTERVENTIONS:
Procedure: Middle ear fluid and urine. — Middle ear fluid and urine collection.

SUMMARY:
The purpose of this epidemiological study is to identify and characterize the bacteria causing Acute Otitis Media episodes in children aged >= 3 months to < 5 years in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Age: >= 3 months and < 5 years at the time of enrolment. The subject becomes ineligible on the fifth birthday.
* Signs, symptoms, and conditions:
* One of the functional or general signs of otalgia, conjunctivitis, fever AND EITHER
* Paradise's criteria, OR
* Spontaneous otorrhoea of less than 1 day.
* Onset of signs and symptoms of acute otitis media within 3 days prior to diagnosis of acute otitis media by a physician. To be included as treatment failure, subjects must have then received antibiotic treatment from the physician, but remain symptomatic 2-3 days after initiation of treatment.
* Written informed consent obtained from parent(s) or Legally Acceptable Representative prior to study start.

Exclusion Criteria:

* Hospitalised during the diagnosis of acute otitis media or during treatment,
* Otitis externa, or otitis media with effusion,
* Presence of a transtympanic aerator,
* Systemic antibiotic treatment received for a disease other than acute otitis media in the 3 days prior to enrolment,
* Receiving antimicrobial prophylaxis for recurrent acute otitis media,
* Provision of antibiotic by the ear nose and throat specialist at the enrolment visit, prior to the sampling of the middle ear fluid by tympanocentesis or spontaneous otorrhoea,
* Patients on antibiotics for acute otitis media who are clinically improving.
* Child in care.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged >= 3 months to < 5 years visiting ear, nose and throat specialists for the treatment of acute otitis media.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of bacterial pathogens isolated from middle ear fluid samples. | 12 Months

SECONDARY OUTCOMES:
Occurrence of bacterial serotypes. | 12 Months
Antimicrobial susceptibility of bacteria isolated from middle ear fluid samples, as assessed by standard microbiological techniques. | 12 Months
Occurrence of treatment failure of acute otitis media and of recurrent acute otitis media. | 12 Months
Occurrence of spontaneous otorrhoea. | 12 Months
Occurrence of bacteria in acute otitis media cases with treatment failure and in new Acute Otitis Media cases without treatment therapy. | 12 Months
Occurrence of bacteria in acute otitis media cases vaccinated with a pneumococcal vaccine. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline